CLINICAL TRIAL: NCT06926686
Title: Prospective Comparison of Acellular Dermal Matrix and Autologous Tarsus for Correction of Lower Eyelid Retraction
Brief Title: Acellular Dermal Matrix vs Autologous Tarsus for Correction of Lower Eyelid Retraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 863946
Record Dates: First submitted 2025-04-11; First posted 2025-04-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-01

CONDITIONS: Lower Eyelid Retraction
Keywords: eyelid malposition

STUDY DESIGN:
Intervention Model Description: Non-masked prospective randomized two-armed interventinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous tarsus (Active Comparator): Surgical implantation to elongate the lower eyelid
  Interventions: Procedure: Autologous tarsus
- A cellular dermal matrix (Permacol) (Active Comparator): Surgical implantation to elongate the lower eyelid
  Interventions: Procedure: Acellular dermal matrix

INTERVENTIONS:
Procedure: Autologous tarsus — Surgical implantation of autologous tarsus to the lower eyelid
  Arms: Autologous tarsus
Procedure: Acellular dermal matrix — Surgical implantation of acellular dermal matrix to the lower eyelid
  Arms: A cellular dermal matrix (Permacol)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two promising implants in treatment of lower eyelid retraction in 40 patients. This condition often resulting from injury, surgical complications, or thyroid eye disease. The main questions it aims to answer are:

Which implant provides better long-term stability of the eyelid malposition?

Does one implant minimize complications and improve patient outcomes more effectively than the other?

This study will compare the use of donor sclera implants to a cellular dermal matrix to see if either offers superior results in terms of reducing graft shrinkage and improving eyelid positioning.

Participants will:

Undergo lower eyelid reconstruction surgery with one of the two implants.

Be monitored for postoperative outcomes, including eyelid position, recurrence rates, and complications over a follow-up period 6 months.

DETAILED DESCRIPTION:
The study aims to find the best way to surgically correct lower eyelid retraction, a condition where the lower eyelid droops, leading to eye dryness, irritation, and potential vision problems. This condition can arise from various causes like thyroid eye disease, complications from eyelid or eye socket surgeries, burns, or injuries. The goal of the study is to determine which "spacer" graft works best to lift the eyelid back into its correct position and provide long-lasting results.

Currently, there's no universally agreed-upon optimal spacer-graft for this condition. Surgeons at the department of Ophthalmology at Haukeland University Hospital are conducting a study to compare two promising spacer graft materials: acellular dermal matrix (Permacol), a processed tissue that encourages tissue regeneration, and autologous tarsus, tissue taken from the patient's own upper eyelid.

Forty patients needing surgery for lower eyelid retraction will be inculded in this study. They will be randomly assigned to receive either the Permacol graft or the autologous tarsus graft. The surgical procedure involves making an incision inside the lower eyelid, separating the retractors (muscles that pull the eyelid down), and inserting the chosen spacer graft between the tarsus (the eyelid's supporting structure) and the retractors. This lifts the eyelid to the correct position.

Patients will be followed up for six months after surgery. Doctors will measure the position of the eyelid, how well the eye closes, and signs of dryness or damage to the eye surface. Patients will also be asked about pain/discomfort, and satisfaction with the cosmetic outcome. The study will track any complications, such as infection or recurrence of the eyelid retraction.

The study will compare the two groups to see which graft provides better eyelid positioning, reduces symptoms, and has fewer complications. Statistical analysis will be used to determine if there are significant differences between the two treatment groups.

The results of this study will provide valuable information for surgeons treating lower eyelid retraction, helping them choose the most effective and safe graft material for their patients. The procedures will be performed by experienced surgeons at Haukeland University Hospital, ensuring patient safety. The study adheres to ethical guidelines, and patients will provide informed consent before participating.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-75 years.
* Grade 2 or higher lower eyelid retraction (according to the retraction grading scale).
* Candidate for surgical correction due to functional or cosmetic reasons.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Active ocular or eyelid infection.
* History of severe scarring or keloid formation.
* Concurrent orbital or eyelid malignancies. Pregnancy or lactation. Uncontrolled systemic diseases (e.g., diabetes, immune disorders). Previous eyelid surgery on the affected eye.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Medial reflex distance 2 | From baseline to 6 months follow-up.
  Number of patients with ≥ 1 mm reduction in medial reflex distance 2

SECONDARY OUTCOMES:
Vertical eyelid aperture | From baseline to 6 months follow-up.
  Number of patients with ≥ 1 mm reduction in vertical eyelid aperture
Scleral show | From baseline to 6 months follow-up.
  Number of patients with ≥ 1 mm reduction in scleral show
  .
Lagophthalmos | From baseline to 6 months follow-up.
  Number of patients with ≥ 1 mm reduction in lagophthalmos
  .
Oxford staining scale | From baseline to 6 months follow-up.
  Number of patients with ≥ 1 reduction in Oxford staining scale (objective assessment of keratopathy). Oxford staining scale range from 0-4, and a higher score mean a worse outcome.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Hans Olav Ueland, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vetslandet, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study group because concent is not obtained to share personal data.

REFERENCES:
- [Result] Ferri M, Oestreicher JH. Treatment of post-blepharoplasty lower lid retraction by free tarsoconjunctival grafting. Orbit. 2002 Dec;21(4):281-8. doi: 10.1076/orbi.21.4.281.8555. PMID 12610767
- [Result] Tao JP, Aakalu VK, Wladis EJ, Sobel RK, Freitag SK, Foster JA, Yen MT. Bioengineered Acellular Dermal Matrix Spacer Grafts for Lower Eyelid Retraction Repair: A Report by the American Academy of Ophthalmology. Ophthalmology. 2020 May;127(5):689-695. doi: 10.1016/j.ophtha.2019.11.011. Epub 2019 Dec 30. PMID 31899031
- [Result] Park E, Lewis K, Alghoul MS. Comparison of Efficacy and Complications Among Various Spacer Grafts in the Treatment of Lower Eyelid Retraction: A Systematic Review. Aesthet Surg J. 2017 Jul 1;37(7):743-754. doi: 10.1093/asj/sjx003. PMID 28333254
- [Result] Zucal I, Waldner M, Shojaati G, Schweizer R, Klein HJ, Giovanoli P, Plock JA. Burn Scar Ectropion Correction: Surgical Technique for Functional Outcomes. Ann Plast Surg. 2022 Mar 1;88(3):271-276. doi: 10.1097/SAP.0000000000003047. PMID 35130205
- [Result] Osaki TH, Monteiro LG, Osaki MH. Management of eyelid retraction related to thyroid eye disease. Taiwan J Ophthalmol. 2022 Feb 14;12(1):12-21. doi: 10.4103/tjo.tjo_57_21. eCollection 2022 Jan-Mar. PMID 35399960